CLINICAL TRIAL: NCT05465811
Title: Effects of Telerehabilitation on Physical and Mental Health of the Elderly in the Covid-19 Pandemic Context: A Pilot Study
Brief Title: Telerehabilitation on Physical and Mental Health of the Elderly in the Covid-19 Pandemic Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Assistant Professor, Paulista University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54143121.1.0000.5402
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Elderly Women
Keywords: Health Services for the Aged; Telemonitoring; Exercise; Health Education; COVID-19
MeSH Terms: conditions — Motor Activity; Health Education; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Experimental): Before the intervention period, the following tests will be applied: SARC-F, Short Physical Performance Battery, hand-grip dynamometry, Geriatric Anxiety Inventory, Geriatric Depression Scale and Pittsburgh Sleep Quality Index.
  Interventions: Other: Program of physical exercises and health education by telerehabilitation
- Follow-up (Experimental): After the intervention period, the following tests will be applied: SARC-F, Short Physical Performance Battery, hand-grip dynamometry, Geriatric Anxiety Inventory, Geriatric Depression Scale and Pittsburgh Sleep Quality Index.
  Interventions: Other: Program of physical exercises and health education by telerehabilitation

INTERVENTIONS:
Other: Program of physical exercises and health education by telerehabilitation — To carry out the telerehabilitation program, the Google Meet platform will be used in order to provide the synchronous service model. This will occur for a period of 16 weeks, three weekly sessions lasting 50 minutes, (total of 48 sessions). The sessions will be given by physiotherapists and students in their final year of graduation in physiotherapy, which will consist of the following phases: initial rest, warm-up, resistance exercises, stretching exercises, relaxation and final rest.
  In addition, in exchange for the warm-up phase, every 12 sessions, the telerehabilitation program also will have an approach through health education, using presentations, digital booklets and direct conversation between therapist and participants. The themes exhibited (importance of physical exercise in the pandemic context, reduction of the risk of falls through changes in the home environment and physiological changes resulting from aging) will intend to make them aware of better lifestyle habits.

SUMMARY:
Introduction: Due to the COVID-19 pandemic scenario, social distancing has become the main strategy to contain this pandemic, causing negative impacts on the physical and mental health of the elderly population. To promote the continuity of offering health services during isolation telerehabilitation was used. Thus, it is important to investigate the effect of a physical exercise program and health education through telerehabilitation on physical and mental aspects in order to establish it as an alternative care for the elderly. Objectives: To evaluate the effect of a program of physical exercises and health education by telerehabilitation on signs of sarcopenia, physical performance, hand grip strength and levels of anxiety, depression and sleep quality in elderly women. Method: In this non-randomized clinical trial, considered a pilot study, eight elderly women (73,00±4,69 years old) will be submitted to 16 weeks of intervention through a program of physical exercise and health education using the Google Meet platform (synchronous online), frequency of 3 weekly sessions and duration of 50' (Initial rest: 5'; Warm-up: 15': Resistance exercises: 20'; Stretching exercises: 5'; Relaxation and final rest: 5'). Before and after the intervention period, the following tests will be applied: SARC-F, Short Physical Performance Battery, hand-grip dynamometry, Geriatric Anxiety Inventory, Geriatric Depression Scale and Pittsburgh Sleep Quality Index. To compare the two moments, the paired Student's T-test or Wilcoxon test (normality assessed by the Shapiro-Wilk test) will be used with p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60 years or older;
* Able to perform all the proposed assessments;
* Not present cognitive impairment according to the assessment of mental status through the Mini Mental State Examination;
* Participate in the supervised physical exercise program in person, prior to the beginning of the COVID-19 pandemic.

Exclusion Criteria:

* had a frequency of participation in the program below 75%.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Signs of sarcopenia | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  Sarcopenia will identify and track by the SARC-F questionnaire, composed of five self-reported questions, based on muscle strength activities, ambulation, rising from a chair, climbing stairs and history of falls, in combination with measurement of the right calf circumference as an indirect assessment of muscle mass.
  The total score will obtain by means of the sum of the questions (maximum 2 points for each) and the measurement of calf circumference (women: > 33 cm = 0; ≤ 33cm =10 points). This questionnaire is valid for Portuguese Language since 2016.
Physical Performance | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  Physical performance will be evaluated using the SPPB, a simple tool that can help to track the risk of falls by identifying risk factors related to the assessed domains.
  This tool has three domains: static balance, lower limbs strength and gait speed. The total SPPB score is made by adding these three domains and can vary between 0 and 12 points.
Hand Grip Strength | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  Hand grip strength will be assessed using a manual dynamometer (Crown produced by the industrial technique Oswaldo Filizola Ltda) with a capacity of 50 kilograms-force, following the protocol proposed by Robert et al.
  During the test, the participant remains seated with the forearms resting on the arms of the chair with wrists in a neutral position and her thumbs facing up. The evaluator assists by holding the base of the dynamometer in the palm of the hand in order to nullify the effect of gravity on the test, while the participant holds the dynamometer. In this way, the patient is asked to press as long and strong as possible or until the pointer stops rising. The test is performed three times in each hand, alternating between them, with an interval of 20 seconds for each attempt. The value recorded regarding strength was the highest among the six measures.
Anxiety symptoms | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  The GAI is an instrument designed to assess anxiety symptoms in elderly individuals, with viable application in situations of fatigue, low educational level or mild cognitive impairment.
  The inventory consists of 20 items with dichotomous responses, with a cut-off point of 10/11 for the detection of generalized anxiety disorder. The GAI will be translated and adapted into Brazilian Portuguese, called the Geriatric Anxiety Inventory (GAI-BR), contributing to a quick, effective and low-cost evaluation with satisfactory validity.
Depressive symptoms | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  The GDS-15 is a self-assessment scale that analyzes the presence of suspected depression in the elderly, easy to apply and low cost. Its reduced version consists of 15 questions, with dichotomous answers (yes/no), in which 0 points are scored when the answer is different from the example in parentheses and 1 point when the answer is the same as the example in parentheses. A 5-point cut-off for the GDS-15 indicates the presence of suspected depression.
Sleep quality | This outcome will be evaluated in two different moments. The first evaluation will be performed at baseline and the second evaluation will be perfomed after 16 weeks of telerehabilitation (follow-up)
  The PSQI is a questionnaire composed of 21 items that assesses subjective quality of sleep and disorders over the last month, in which 19 questions are self-assessment and 5 questions that must be answered by bedmates or roommates.
  The PSQI analyzes seven issues: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disorders, use of sleeping medications, and daytime dysfunction. Its score ranges from 0 to 21 and indicates the overall quality of sleep, classifying individuals into good sleep quality (score less than 5) and poor sleep quality (score greater than 5), that is, the lower the score, the better the sleep quality score.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided